CLINICAL TRIAL: NCT04778007
Title: Validity and Reliability of the Turkish Version of the Laryngopharyngeal Measure of Perceived Sensation Questionnaire
Brief Title: The Validation of the Turkish Version of the LUMP Questionnaire
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Yavuz Atar, Assoc. Prof., M.D., Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 90
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Globus Pharyngeus; Validation
Keywords: globus; sensation; pharyngeus; laryngopharyngeal; measure; perceived; Turkish
MeSH Terms: conditions — Globus Sensation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Globus pharyngeus patients: The first group consists of 80 globus pharyngeus patients who have at least a year of globus sensation complaints. The participants will given the Turkish Version of the Laryngopharyngeal Measure of Perceived Sensation Questionnaire (T-LUMP), consist of 8 questions, Glasgow Edinburg Throat Scale, and Visual analog scale. After the two weeks, 80 participants will given the T-LUMP and Visual analog scale for sampling.
  Interventions: Other: Turkish Version of Laryngopharyngeal Measure of Perceived Sensation Questionnaire
- Healty subjects: The second group consists of 80 healty participants will given the T-LUMP consist of 8 questions, Glasgow Edinburg Throat Scale, and Visual analog scale
  Interventions: Other: Turkish Version of Laryngopharyngeal Measure of Perceived Sensation Questionnaire

INTERVENTIONS:
Other: Turkish Version of Laryngopharyngeal Measure of Perceived Sensation Questionnaire — The Turkish Version of Laryngopharyngeal Measure of Perceived Sensation Questionnaire consists of 8 questions related with globus pharyngeus symptoms.

SUMMARY:
Purpose of the study is the validity and reliability of the Turkish version of the Laryngopharyngeal Measure of Perceived Sensation (T-LUMP) Questionnaire, so that it would be used as an assessment tool for Turkish globus pharyngeus patients.

DETAILED DESCRIPTION:
Globus pharyngeus or sensation may be defined as a feeling of something a lump in the throat without dysphagia. The study will assess the construct validity and reliability of the Turkish version of Laryngopharyngeal Measure of Perceived Sensation (T-LUMP) Questionnaire. The investigators developed the Turkish version of this questionnaire (T-LUMP), according to the cross-cultural adaptation guidelines. Two translators translated the LUMP into Turkish and a native English language speaker reverse-translated it into English. The back translation was sent to the original author for proofreading. The final version of the LUMP questionnaire consisted of 8 basic and understandable questions related with globus pharyngeus symptoms.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with globus pharyngeus in study group
* Able to speak, read, understand and write in Turkish
* give a consent form

Exclusion Criteria:

* patients with dysphagia or odynophagia
* laryngeal organic pathologies
* pharyngeal organic pathologies
* epiglottic retroversion
* malignancy
* pregnancy
* mental disorders
* neurological disorders
* major psychiatric disorders
* Underwent laryngectomy/neck dissection/tracheostomy/neck radiotherapy
* Underwent any surgery last a year
* Cognitive limitations
* give not a consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who diagnosed with Globus pharyngeus
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The outcomes of the Turkish Version of Laryngopharyngeal Measure of Perceived Sensation Questionnaire | Baseline
  Turkish version of the questionnaire consists of 8 questions about globus pharyngeus consequences during patients at least a year and healty subjects. The minimum score is 0 and maximum score is 32. The lower scores mean no problem, higher scores mean significant problem.
The outcomes of the Turkish Version of Laryngopharyngeal Measure of Perceived Sensation Questionnaire | 2 weeks
  Turkish version of the questionnaire consists of 8 questions about globus pharyngeus consequences during patients at least a year. The minimum score is 0 and maximum score is 32. The lower scores mean no problem, higher scores mean significant problem.
The outcomes of Glasgow Edinburg Throat Scale | Baseline
  It was assessed by Turkish validated Glasgow Edinburg Throat Scale that a self questionnaire in globus pharyngeus patients. The minimum score is 0 and maximum score is 7 per question. The high scores were worst low scores were good.
The outcomes of the visual analog scale | Baseline
  The globus sense was assessed by visual analog scale. The minimum score is 0 and maximum score is 100 on a line as 100 millimetres . The high scores were worst low scores were good.
The outcomes of the visual analog scale | 2 weeks
  The globus sense was assessed by visual analog scale. The minimum score is 0 and maximum score is 100 on a line as 100 millimetres . The high scores were worst low scores were good.

SECONDARY OUTCOMES:
Eating Assessment Tool | Baseline
  The Turkish validated questionnaire consists of 10 questions that scores are from 0 to 40. Low score is better, higher score is worse.
Penetration and aspiration scale | Baseline
  The scale consists of 8 levels for assessment of penetration and aspiration. The scores are from 0 to 8. Low score is better, higher score is worse.
Yale pharyngeal residue severity rating scale | Baseline
  The scale consists of 5 assessment units for pharyngeal residue. The scores are from 1 to 5. Low score is better, higher score is worse.

OTHER OUTCOMES:
Subject demographics | Baseline
  The median values of age and ratio of gender, and education with profession profile in all groups

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Atar, Asso.Prof,MD, Study Chair — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Yavuz Atar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melancon CC, Russell GB, Ruckart K, Persia S, Peterson M, Carter Wright S Jr,, Madden LL. The development and validation of the laryngopharyngeal measure of perceived sensation. Laryngoscope. 2020 Dec;130(12):2767-2772. doi: 10.1002/lary.28348. Epub 2019 Oct 23. PMID 31643076
- [Background] Korkmaz MO, Tuzuner A, Bahcecitapar M, Karacaer C. Reliability and Validity of the Turkish Version of the Glasgow-Edinburgh Throat Scale: Use for a Symptom Scale of Globus Sensation in Turkish Population. Turk Arch Otorhinolaryngol. 2020 Mar;58(1):41-47. doi: 10.5152/tao.2020.4686. Epub 2019 Aug 15. PMID 32313894